CLINICAL TRIAL: NCT02090140
Title: Randomized Controlled Trial of Microfracture Versus Adipose Derived Stem Cells for the Treatment of Isolated Articular Cartilage Defects
Brief Title: Microfracture Versus Adipose Derived Stem Cells for the Treatment of Articular Cartilage Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Kentucky (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-2838
Record Dates: First submitted 2014-03-11; First posted 2014-03-18 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Lesion of Articular Cartilage of Knee
Keywords: cartilage/transplantation; cartilage, articular/injuries; cartilage, articular/surgery; chondrocytes/cytology; knee injuries/surgery; knee joint/surgery; orthopedic procedures/methods; tissue engineering; tissue scaffolds; arthroscopy/methods; chondrocytes/transplantation; adipose tissue/cytology; cartilage, articular/cytology; chondrogenesis/physiology; osteogenesis/physiology; stem cell transplantation/methods; stem cells; tissue engineering/methods; cartilage, articular/pathology; chondrocytes/pathology; knee joint/pathology; platelet-rich plasma
MeSH Terms: conditions — Wounds and Injuries; Knee Injuries | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADSC Application (Experimental): Patients undergo an arthroscopic surgical procedure, ADSC application, followed by physical therapy.
  Interventions: Procedure: ADSC Application
- Microfracture Arm (Active Comparator): Patients undergo an arthroscopic surgical procedure, microfracture, followed by physical therapy.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: ADSC Application — Patients will undergo arthroscopic resection of approximately 5cc of the infrapatellar fat pad, which will be collected for processing for a population of ADSCs. Patients will undergo arthroscopy and preparation of the chondral defect and removal of the calcified cartilage layer. Tisseel Fibrin glue will be placed at the base of the defect side, followed by the application of the acellular collagen dermal matrix, ADSCs, and an additional layer of fibrin glue.
  Arms: ADSC Application
Procedure: Microfracture — Microfracture surgery is the standard of care for articular cartilage lesions. Patients will undergo arthroscopy with standard technique of microfracture preparation, including the creation of vertical, stable defect edges and removal of the calcified cartilage layer. A microfracture awl will then be used to perform the microfracture technique (6mm below the subchondral plate).
  Arms: Microfracture Arm

SUMMARY:
The purpose of this study is to compare two biologic methods for the treatment of articular cartilage defects in the knee. The first method, microfracture, is the standard of care and is routinely used to recruit cells from the subchondral bone marrow to the site of cartilage loss. The second method is the application of adipose-derived stem cells (ADSCs) to the defect site. In theory, ADSCs on a collagen scaffold should enable the delivery of more specific progenitor cells to the site of injury, resulting in better regeneration and integration of articular cartilage at the site of a defect as compared to the microfracture method.

DETAILED DESCRIPTION:
Patients enrolled in the ADSC cohort will undergo the following procedures: arthroscopic resection of approximately 5cc of the infrapatellar fat pad using a motorized shaver (standard use in arthroscopy). Fat will be collected in a sterile Aquavage Collection System (AV1200, MD Resources, Livermore, CA) and kept sealed until processing. Fat will then immediately be processed in the Harvest Adiprep System to separate a population of ADSCs. This system concentrates an average of 5 x 105 cells/ml. All specimens will be processed using routine sterile procedures within the operating room; cells destined for implantation will not leave the operating room. Concurrently, patients will undergo arthroscopy and similar preparation of the chondral defect and removal of the calcified cartilage layer. However, no puncture of the subchondral bone will be performed. A layer of fibrin glue (Tisseel) will be placed at the base of the defect to seal off any bleeding from the subchondral plate followed by the application of the acellular dermal matrix (Allopatch HD, MTF Corporation, Edison, NJ, USA)and ADSCs. An additional layer of Tisseel will then be applied over the cells and matrix. No additional fixation will be applied. The matrix and cells will be recessed below the articular surface by an average of 1mm.

They will then complete outcome questionnaires and additional MRI scans at 6, 12, and 24 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Must be between ages 18 and 50 years.
* Must have a discrete, contained chondral defect less than 400mm^2 located on the medial or lateral femoral condyle
* Must have overall neutral lower limb mechanical alignment (<5 degrees varus or valgus).

Exclusion Criteria:

* Ages younger than 18 years and older than 50 years.
* If they have undergone previous chondral procedures
* If they have pre-existing osteoarthritis (Kellegren-Lawrence Grade ≥2)
* If they have a BMI >30.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health Scores on the KOOS Questionnaire | Completed at baseline, 6 months, 12 months, and 24 months post-operatively.
  The Knee Osteoarthritis Outcome Score (KOOS), a standard outcome questionnaire for the assessment of health-related quality of life, will be completed.

SECONDARY OUTCOMES:
Activity Level on the Tegner Activity Scale | Completed at baseline, 6 months, 12 months, and 24 months post-operatively.
  The Tegner Activity scale, a standard outcome questionnaire for assessment of activity levels, will be completed.
Cartilage Composition Assessment by MRI Scan | Assessed at baseline, 6 months, 12 months, and 24 months post-operatively.
  Magnetic resonance imaging scans consisting of routine clinical sequences and T2 and T1p quantitative maps will be conducted. T1p and T2 mapping will be used to assess regenerative cartilage composition compared to surrounding normal cartilage, surface integrity, average cartilage thickness, and the percentage to which the defect is filled.
Functionality Scores on the Lysholm Scale | Completed at baseline, 6 months, 12 months, and 24 months post-operatively.
  The Lysholm Scale, a standard outcome questionnaire for assessment of knee functionality, will be completed.
Pain Scores on the Visual Analog Scale (VAS) | Completed at baseline, 6 months, 12 months, and 24 months post-operatively.
  The Visual Analog Scale, a standard outcome questionnaire for assessment of pain levels, will be completed.
Health Scores on Veterans-Rand (VR-12) Survey | Completed at baseline, 6 months, 12 months, and 24 months post-operatively.
  The Veterans-Rand survey, a standard outcome questionnaire for assessment of health and quality of life, will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dragoo, MD, Principal Investigator — University of Colorado, Denver; Seth L Sherman, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford Medical Outpatient Center, Redwood City, California
  - Kerlan Jobe Orthopedic Institute, Santa Monica, California
  - UC Health Steadman Hawkins Clinic - Denver Inverness, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedi A, Feeley BT, Williams RJ 3rd. Management of articular cartilage defects of the knee. J Bone Joint Surg Am. 2010 Apr;92(4):994-1009. doi: 10.2106/JBJS.I.00895. PMID 20360528
- [Background] Knutsen G, Engebretsen L, Ludvigsen TC, Drogset JO, Grontvedt T, Solheim E, Strand T, Roberts S, Isaksen V, Johansen O. Autologous chondrocyte implantation compared with microfracture in the knee. A randomized trial. J Bone Joint Surg Am. 2004 Mar;86(3):455-64. doi: 10.2106/00004623-200403000-00001. PMID 14996869
- [Background] Dragoo JL, Samimi B, Zhu M, Hame SL, Thomas BJ, Lieberman JR, Hedrick MH, Benhaim P. Tissue-engineered cartilage and bone using stem cells from human infrapatellar fat pads. J Bone Joint Surg Br. 2003 Jul;85(5):740-7. PMID 12892203
- [Background] English A, Jones EA, Corscadden D, Henshaw K, Chapman T, Emery P, McGonagle D. A comparative assessment of cartilage and joint fat pad as a potential source of cells for autologous therapy development in knee osteoarthritis. Rheumatology (Oxford). 2007 Nov;46(11):1676-83. doi: 10.1093/rheumatology/kem217. Epub 2007 Sep 26. PMID 17901063
- [Background] Koh YG, Choi YJ. Infrapatellar fat pad-derived mesenchymal stem cell therapy for knee osteoarthritis. Knee. 2012 Dec;19(6):902-7. doi: 10.1016/j.knee.2012.04.001. Epub 2012 May 14. PMID 22583627
- [Background] Ma A, Jiang L, Song L, Hu Y, Dun H, Daloze P, Yu Y, Jiang J, Zafarullah M, Chen H. Reconstruction of cartilage with clonal mesenchymal stem cell-acellular dermal matrix in cartilage defect model in nonhuman primates. Int Immunopharmacol. 2013 Jul;16(3):399-408. doi: 10.1016/j.intimp.2013.02.005. Epub 2013 Mar 13. PMID 23499511
- [Background] Giavaresi G, Bondioli E, Melandri D, Giardino R, Tschon M, Torricelli P, Cenacchi G, Rotini R, Castagna A, Veronesi F, Pagani S, Fini M. Response of human chondrocytes and mesenchymal stromal cells to a decellularized human dermis. BMC Musculoskelet Disord. 2013 Jan 7;14:12. doi: 10.1186/1471-2474-14-12. PMID 23294867
- [Background] Desando G, Cavallo C, Sartoni F, Martini L, Parrilli A, Veronesi F, Fini M, Giardino R, Facchini A, Grigolo B. Intra-articular delivery of adipose derived stromal cells attenuates osteoarthritis progression in an experimental rabbit model. Arthritis Res Ther. 2013 Jan 29;15(1):R22. doi: 10.1186/ar4156. PMID 23360790
- [Background] Koh YG, Jo SB, Kwon OR, Suh DS, Lee SW, Park SH, Choi YJ. Mesenchymal stem cell injections improve symptoms of knee osteoarthritis. Arthroscopy. 2013 Apr;29(4):748-55. doi: 10.1016/j.arthro.2012.11.017. Epub 2013 Jan 29. PMID 23375182
- [Background] Wickham MQ, Erickson GR, Gimble JM, Vail TP, Guilak F. Multipotent stromal cells derived from the infrapatellar fat pad of the knee. Clin Orthop Relat Res. 2003 Jul;(412):196-212. doi: 10.1097/01.blo.0000072467.53786.ca. PMID 12838072